CLINICAL TRIAL: NCT03896620
Title: Recognition of Circulating Tumor DNA in Soft Tissue Sarcoma
Status: Recruiting | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Ciani M Ellison, MD, Assistant Professor, Medical College of Wisconsin
Other Study IDs: PRO00034441
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Sarcoma
Keywords: Sarcoma; ctDNA
MeSH Terms: conditions — Sarcoma | interventions — Postoperative Period; Drug Therapy; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — In this project, the investigator will do genetic testing on blood and tumor samples. Whole genome sequencing will be included as part of the genetic testing for this research. Genetic testing will be done because the study doctor would like to identify new biomarkers of sarcoma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Stage II-III Sarcomas undergoing preoperative radiation therapy (RT): This group will have preoperative chemotherapy (if administered), preoperative radiation and surgery.
  Interventions: Device: Preoperative RT; Drug: Chemotherapy; Other: Surgery
- Stage II-III Sarcomas undergoing postoperative RT: This group will have surgery, postoperative radiation, post operative chemotherapy (if administered).
  Interventions: Device: Postoperative RT; Drug: Chemotherapy; Other: Surgery
- Stage IV Sarcomas: This group will only have chemotherapy.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Device: Preoperative RT — Radiation delivered before surgery.
  Groups: Stage II-III Sarcomas undergoing preoperative radiation therapy (RT)
Device: Postoperative RT — Radiation delivered after surgery.
  Groups: Stage II-III Sarcomas undergoing postoperative RT
Drug: Chemotherapy — Physician's choice of chemotherapy.
Other: Surgery — Surgical excision of tumor.
  Groups: Stage II-III Sarcomas undergoing postoperative RT; Stage II-III Sarcomas undergoing preoperative radiation therapy (RT)

SUMMARY:
A tissue biopsy is currently the only clinical test or procedure that is able to confirm the initial diagnosis of soft tissue or metastatic sarcoma and evaluate its progress during treatment. However, tissue biopsy collection can be challenging (depending on the location of the tumor), and this procedure poses physical risks to the patient. A tissue biopsy also needs to be recollected at various time points in order to assess if the patient is responding to treatment.

In this project, the investigator would like to collect blood samples in addition to the sample of the tumor that will be collected before treatment is started. The investigator would like to analyze both blood and tumor, in hopes of identifying new biomarkers of sarcoma that can help the study doctors better diagnose sarcoma for patients in the future without needing to collect a piece of their tumor.

A biomarker is something found in the blood, other body fluids, or tissues that can be used to measure the progress of disease, how a treatment is working, or its likelihood of being successful. In this project, the investigator would like to compare ctDNA from blood to the DNA in the tumor. ctDNA, or circulating tumor DNA, is DNA originating from the tumor that is present in the blood. It can be assessed by taking an additional sample of blood when it will be collected for normal laboratory tests. These biomarkers may also help the study doctors detect how a patient is responding to their treatment or help predict their response to future treatment.

DETAILED DESCRIPTION:
In the proposed study, the investigators wish to prospectively collect blood samples from 25 patients with localized soft tissue sarcomas and 25 patients with metastatic sarcoma (schema III) at various time points outlined. The presence/absence, as well as the change of ctDNA in circulation, will then be measured after the therapies administered and correlated with overall survival, progression-free survival and local control.

The risks to the subjects enrolled on this study include the general risks of undergoing the standard procedures, such as blood draws, imaging, radiation therapy, chemotherapy and surgery, which will be discussed prior to the therapies and images each patient undergoes. The risks of the procedures are not risks of the study with exception to blood draws. There is also a risk of loss of confidentiality, but the data will be deidentified once acquired. Thus, this risk is minimal.

ELIGIBILITY:
Inclusion Criteria:

* Have signed an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved informed consent form (ICF) prior to any study-specific evaluation.
* Diagnosis of soft tissue sarcoma.
* ≥ 18 years of age.
* Planned biopsy obtained within four weeks after registration.
* History and physical within eight weeks prior to registration.
* For stage II-III patients, no prior therapy to primary site of sarcoma.
* Computerized tomography (CT), positron emission tomography (PET) /CT or MR imaging of the affected primary site obtained in stage II-III or metastatic site in stage IV patients within eight weeks prior to registration.
* CT chest or PET /CT acquired to assess distant disease within eight weeks prior to registration for stage II-III patients.
* Karnofsky Performance Scale (KPS) 60 or above within four weeks prior to registration.
* Documentation of stage within eight weeks prior to registration.
* Biopsy of primary or metastatic disease site must be safe, feasible and in concordance with standard of care per the treating physician and/or radiologist.
* Life expectancy ≥ 12 weeks.

Exclusion Criteria:

* Pregnant women.
* Patients with a history of metastatic disease from a primary other than sarcoma.
* Patients who cannot undergo imaging as part of treatment planning or surveillance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with localized, stage II-III or stage IV histologically confirmed soft tissue sarcomas of the extremity, chest wall or retroperitoneal primaries will be eligible for this study. Stage IV patients may have had prior therapy but must obtain a biopsy within registration requirements for study enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-06-18 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
ctDNA measure | Reported at baseline, at 4 weeks after first intervention, 4 weeks following radiation treatment, 4 weeks post third intervention, 1 year.
  Blood samples will be collected. ctDNA is measured in percentage: variant allele fraction percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Meena Bedi, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No